CLINICAL TRIAL: NCT07137949
Title: Delirium in Neurodegenerative Disease Patients: A Music Therapy Intervention for Hospital Care
Acronym: DyNamic
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-46190
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Delirium
Keywords: Music therapy; Hospital acquired delirium; Neurodegenerative disease patients
MeSH Terms: conditions — Delirium | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music therapy (Experimental): Participants will undergo one-on-one music therapy (MT) sessions of approximately 30 minutes duration conducted by a board-certified music therapist. Sessions will be customized to address patient needs but will consistently adhere to the four principal MT methods of re-creation, composition, improvisation, and therapeutic listening experiences.
  Interventions: Behavioral: Music therapy

INTERVENTIONS:
Behavioral: Music therapy — Live music therapy (MT) sessions will occur 3 times/week, up to 5 sessions. Sessions will be responsive to patient preferences, culture, and identity using information gained from medical record review, intake assessment, and in the moment therapeutic assessments.

SUMMARY:
In this pilot study a new kind of music therapy will be created and tested to help prevent confusion, called delirium, that can happen in the hospital. This can affect people with brain diseases like Alzheimer's disease and Parkinson's disease.

Each of the anticipated 30 participants will have up to five music therapy sessions. The sessions will be made just for them and may include live music, playing instruments, or listening to recorded music. Surveys will be used to learn how easy the therapy is to do in the hospital and what people think about how helpful the sessions may be for future patients.

ELIGIBILITY:
Inclusion Criteria:

* Admitted as inpatient to Boston Medical Center.
* Cognitive impairment or neurodegenerative diseases as defined by either:

  * Diagnosis of Parkinson's Disease, Dementia with Lewy Bodies (ICD-10 G20 and G31.83 respectively), Alzheimer's Disease-related dementias (ICD-10 6D80), vascular dementia (F01), or other cognitive impairment (R41) on active problem list or past medical history
  * "Cognitive impairment" on active problem list or past medical history
  * Documentation elsewhere in the electronic medical record (e.g. notes) of any of these conditions
* Participants with cognitive impairment will be included. If unable to consent, legally authorized representative (LAR) based on HRP-013-SOP-LARs, Children, and Guardians will be contacted to consent.
* Spanish speaking participants will be included. Screening and informed consent procedures will be conducted using a certified medical interpreter. All intervention sessions and study team interactions will be conducted using these interpreter services.
* Patients admitted to an intensive care unit will be included as long as they are not receiving continuous intravenous sedative medications. Potential participants in the intensive care unit setting will be discussed with a PI/co-I to ensure participation is appropriate on a case-by-case basis. The PI/Co-I will confirm with the treating physician that there are no reasons as to why the potential participant should not be enrolled in the study.

Exclusion Criteria:

* Admitted to observation status (as these patients would not be expected to remain inpatient long enough to undergo the MT intervention)
* Patients who will be discharged within 24 hours of eligibility based on discussion with primary admitting team
* Self-reported history of musicogenic seizures
* Hearing loss: unable to hear a recorded sound <70 decibels (dB)
* Dislike of music: Barcelona Music Reward Questionnaire score of <40
* Patients who are currently prisoners
* Patients in the intensive care unit receiving continuous intravenous sedative medication
* Pregnant women

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Delirium scores | every 24 hours until discharge (on average 7 days)
  The 3-Minute Diagnostic Interview for the Confusion Assessment Method (3D-CAM) will be used to assess presence and severity of delirium. For participants who cannot complete the 3D-CAM due to non-verbal status, the CAM-ICU will be used in its place.
Number of music therapy sessions successfully completed | during hospitalization, on average 7 days

SECONDARY OUTCOMES:
Number of days that participants screen CAM-positive | during hospitalization, on average 7 days
  The 3-Minute Diagnostic Interview for the Confusion Assessment Method (CAM) will be used to assess delirium. It will provide a binary outcome: delirium present (CAM positive) or absent (CAM negative).
Number of participants given antipsychotic medications | during hospitalization, on average 7 days
  Based on data from the electronic medical record.
Number of participants requiring physical restraints | during hospitalization, on average 7 days
  Based on data from the electronic medical record.
Number of participants with one-to-one sitter orders | during hospitalization, on average 7 days
  Based on data from the electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Kara M Smith, MD MSCI FAAN, Principal Investigator — Boston Medical Center, Neurology
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No